CLINICAL TRIAL: NCT03225482
Title: Cognitive Rehabilitation for Older Veterans With Mild Cognitive Impairment
Brief Title: Cognitive Rehabilitation Therapy for Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Portland VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NURD-019-16F; I01CX001592 (NIH)
Record Dates: First submitted 2017-07-07; First posted 2017-07-21 (Actual); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Cognitive rehabilitation; Cognitive training; Cognitive remediation
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Two group randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blind to treatment group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ME-CCT (Experimental): 8-week Motivationally Enhanced Compensatory Cognitive Training group
  Interventions: Behavioral: Motivationally Enhanced Compensatory Cognitive Training
- SC (Active Comparator): 8-week Goal-focused Supportive Contact group
  Interventions: Behavioral: Goal-focused Supportive Contact

INTERVENTIONS:
Behavioral: Motivationally Enhanced Compensatory Cognitive Training — ME-CCT is a manualized group-based behavioral intervention (8 weeks, 2 hours per week, 20 hours total) designed to improve cognitive and everyday functioning in patients with MCI.
  Other Names: ME-CCT
  Arms: ME-CCT
Behavioral: Goal-focused Supportive Contact — SC is a group therapy intervention that provides the same frequency and amount of therapist and other group member contact as ME-CCT, but does not provide training in cognitive strategies, lifestyle strategies, or motivational enhancement. The SC intervention focuses on setting and achieving short or long-term goals.
  Other Names: SC
  Arms: SC

SUMMARY:
The number of older Veterans with Mild Cognitive Impairment (MCI) seeking care within the Veterans Affairs (VA) health care system is increasing and is expected to increase more rapidly as Vietnam era Veterans age. The cognitive effects of MCI and subsequent neurodegenerative disorders can adversely affect a Veteran's ability to function independently and failure to provide appropriate intervention can result in an increased need for healthcare services and VA benefits in the future. The VA currently spends over $19,000 annually per patient to care for Veterans with dementia (Zhu et al., 2009), and delaying the onset of dementia even by one to two years will result in substantial financial savings to the VA and quality of life gains for the Veteran. Since present pharmacological interventions have demonstrated limited efficacy, alternative treatments are needed. Therefore, an evidence-based cognitive training intervention that optimally addresses the needs of older Veterans with MCI is of critical importance to the VA patient care mission.

DETAILED DESCRIPTION:
Due to the aging of the United States population, age-related cognitive problems resulting from Alzheimer's disease and other causes of dementia are increasingly prevalent. Before individuals are diagnosed with dementia, they typically exhibit a period of "mild cognitive impairment" (MCI). Mild cognitive problems associated with MCI frequently impact an individual's ability to perform everyday tasks, including working, independent living, and medication adherence. Veterans are at increased risk of cognitive decline, and the Veterans Healthcare Administration (VA) is now providing health care to surging numbers of older Veterans with MCI who report significant cognitive complaints, difficulties with everyday functioning, and concerns about impending dementia. Despite high patient demand, few cognitive rehabilitation interventions exist that specifically address the needs of older Veterans with MCI that are widely accessible, patient-centered, and evidence-based. To the investigators' knowledge, no randomized controlled trials have been conducted that evaluate the efficacy of manualized, brief and inexpensive, yet comprehensive (multi-modal) cognitive rehabilitation interventions for older Veterans with MCI. Hence, the primary objective of this study is to evaluate the efficacy of Motivationally Enhanced Compensatory Cognitive Training (ME-CCT), a manualized cognitive rehabilitation group treatment for older Veterans with MCI. The study's specific aims are to determine whether ME-CCT is effective for: 1) improving objective cognitive performance and functional capacity, 2) improving subjective cognitive complaints, subjective functioning, and collateral measures of everyday function, and 3) increasing modifiable protective factors (e.g., diet, exercise) associated with reduced risk for MCI. The investigators will also explore mediators and moderators of treatment effects. The overall goal is to evaluate a manualized group treatment for the symptoms of MCI that can be readily implemented in VA treatment settings. The study design makes use of the convergent availability of resources at the two participating VA Healthcare Systems in San Diego, California and Portland, Oregon to conduct a randomized controlled trial of ME-CCT. The study will recruit a sample of 216 Veterans (108 at each site) who meet criteria for MCI. Inclusion criteria will be: 1) Veterans 55 years old or older enrolled at one of the participating VAs who are able to provide informed consent, 2) Independently living, 3) Meet criteria for MCI based on previously published criteria (Petersen, 2004; Petersen, 2011), and 4) Willingness to participate in audio-recorded group sessions. Exclusion criteria will be: 1) Current substance use disorder with less than 30 days abstinence, 2) History of schizophrenia, schizoaffective disorder, or other primary psychotic disorder, 3) History of significant head trauma with loss of consciousness >30 minutes, and 4) Auditory or visual impairments that would prevent ability to participate in the cognitive rehabilitation group. Eligible participants will be randomly assigned to either the ME-CCT or an active control group, Goal-focused Supportive Contact (SC). The SC group will provide the same frequency and amount of therapist and peer contact as ME-CCT, but without specific training in cognitive strategies, lifestyle strategies, or motivational enhancement. 8 2-hour long weekly sessions will be delivered in both conditions. Both groups will undergo evaluations at baseline, 4 weeks (midway through the intervention), 8 weeks (immediately following the end of the intervention), and 21 weeks (3 months after completion of the intervention).

ELIGIBILITY:
Inclusion Criteria:

* Veterans >55 years old enrolled at one of the participating VA sites (VASDHS and VAPORHCS) who are able to provide informed consent
* Independently living
* Meet criteria for MCI based on previously published criteria (see below)
* Willingness to participate in audio-recorded sessions.
* MCI Criteria:

  * Concern about a decline in cognitive functioning expressed by a physician, informant, participant or nurse
  * Cognitive impairment in one or more of the following domains

    * executive function
    * memory
    * attention
    * language or visuospatial abilities
  * Normal or minimal impairment in functional activities
  * Does not meet criteria for dementia

Exclusion Criteria:

* Current substance use disorder with < 30 days abstinence
* History of schizophrenia, schizoaffective disorder, or other primary psychotic disorder
* History of significant brain injury with loss of consciousness > 30 minutes
* Auditory or visual impairments that would prevent ability to participate in the cognitive rehabilitation group or benefit from compensatory strategies

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth W. Twamley, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (2):
- United States (2):
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Portland Health Care System, Portland, OR, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were considered enrolled when they signed the informed consent form. Participants then underwent baseline assessment. Once six participants completed baseline assessments, they were randomized as a group to a condition, revealed to them on the first day of treatment. Some participants exited prior to baseline assessment or after baseline assessment but before randomization or the first day of treatment. Thus, the number initiating treatment differs from the number enrolled.
Groups:
- ME-CCT Group: 8-week Motivationally Enhanced Compensatory Cognitive Training group
- Supportive Contact Control Group: 8-week Goal-focused Supportive Contact group
Period: Overall Study
Arm/Group | ME-CCT Group | Supportive Contact Control Group
Started | 79 | 66
Completed | 76 | 61
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Population: 156 participants completed baseline assessments and will be included in the intent-to-treat analyses. This number differs from the number enrolled (193) and the number who started treatment (145).
Groups:
- Total: Total of all reporting groups
Arm/Group | ME-CCT | Supportive Contact Control Group | Total
Number analyzed (Participants) | 84 | 72 | 156
Age, Continuous [Mean (Standard Deviation); unit: year] | 71.2 (8.2) | 71.8 (7.0) | 71.5 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 72 | 65 | 137
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 66 | 57 | 123
  Unknown or Not Reported | 13 | 9 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 10 | 4 | 14
  White | 60 | 60 | 120
  More than one race | 6 | 4 | 10
  Unknown or Not Reported | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Objective Cognitive Performance Composite z Score
Description: Change in composite z score on the following tests:
  Hopkins Verbal Learning Test-Revised (HVLT-R) Brief Visuospatial Memory Test-Revised (BVMT-R) Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-IV) Digit Span WAIS-IV Coding Delis-Kaplan Executive Function System (D-KEFS) Trails, Number and Letter Sequencing D-KEFS Trails, Number-Letter Switching D-KEFS Color-Word Interference Test, Inhibition and Inhibition-Switching A Z score of 0 represents the sample mean. Higher composite Z scores reflect better performance.
Time Frame: assessed at baseline, 8 weeks, 21 weeks; change from baseline to 21 weeks reported.
Population: 114 participants had useable data at baseline and 21 weeks.
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | ME-CCT | Supportive Contact Control Group
Number analyzed (Participants) | 66 | 48
Z score | .24 (.39) | .14 (.35)

2. Primary Outcome: Change in Functional Capacity Performance Composite z Score
Description: Change in composite z score on the following measures:
  UCSD Performance-Based Skills Assessment-Brief (UPSA-B) Medication Management Ability Assessment (MMAA) Neuropsychological Assessment Battery Daily Living Memory Neuropsychological Assessment Battery Judgment Neuropsychological Assessment Battery Driving Scenes A Z score of 0 represents the sample mean. Higher Z scores reflect better performance.
Time Frame: assessed at baseline, 8 weeks, 21 weeks; change from baseline to 21 weeks reported.
Population: 111 participants had useable data at baseline and 21 weeks.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | ME-CCT | Supportive Contact Control Group
Number analyzed (Participants) | 65 | 46
z-score | .11 (.41) | .17 (.61)

3. Secondary Outcome: Change in Subjective Everyday Functioning Composite Score
Description: Change in average total score across Applied Cognition Executive Function and Applied Cognition General Concerns scales.
  The average total score ranges from 8-40, with higher scores reflecting better subjective cognition.
Time Frame: assessed at baseline, 4 weeks, 8 weeks, 21 weeks; change from baseline to 21 weeks reported.
Population: 121 participants had useable data at baseline and 21 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ME-CCT | Supportive Contact Control Group
Number analyzed (Participants) | 69 | 52
score on a scale | 2.41 (4.76) | .64 (4.46)

4. Secondary Outcome: Change in Everyday Cognition Scale
Description: Change in total score on the Everyday Cognition Scale. Total scores range from 39-195, with higher scores reflecting worse everyday cognition.
Time Frame: assessed at baseline, 4 weeks, 8 weeks, 21 weeks; change from baseline to 21 weeks reported.
Population: 122 participants had useable data at baseline and 21 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ME-CCT | Supportive Contact Control Group
Number analyzed (Participants) | 69 | 53
score on a scale | -.32 (.55) | -.10 (.41)

5. Secondary Outcome: Change in Cognitive Activity Inventory
Description: Change in total score on the Cognitive Activity Inventory. Scores represent hours per month of cognitive activity and range from 0-730 (the number of hours in a month). Higher scores represent more hours of cognitive activity.
Time Frame: assessed at baseline, 4 weeks, 8 weeks, 21 weeks; change from baseline to 21 weeks reported.
Population: 120 participants had useable data at baseline and 21 weeks.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ME-CCT | Supportive Contact Control Group
Number analyzed (Participants) | 68 | 52
hours | 24.37 (245.46) | -26.80 (288.83)

6. Secondary Outcome: Change in CHAMPS Physical Activity Questionnaire for Older Adults
Description: Change in total score on the CHAMPS Physical Activity Questionnaire for Older Adults. The score reflects hours of exercise per week and ranges from 0-168 (the number of hours in one week). Higher scores reflect higher levels of exercise.
Time Frame: assessed at baseline, 4 weeks, 8 weeks, 21 weeks; change from baseline to 21 weeks reported.
Population: 116 participants had useable data at baseline and 21 weeks.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ME-CCT | Supportive Contact Control Group
Number analyzed (Participants) | 64 | 52
hours | -2.02 (9.15) | 1.76 (9.80)

7. Secondary Outcome: Change in Portland Cognitive Strategies Scale
Description: Change in total score on the Portland Cognitive Strategies Scale. Scores reflect use of cognitive strategies and range from 0-60, with higher scores reflecting greater use of cognitive strategies.
Time Frame: assessed at baseline, 4 weeks, 8 weeks, 21 weeks; change from baseline to 21 weeks reported.
Population: 119 participants had useable data at baseline and 21 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ME-CCT | Supportive Contact Control Group
Number analyzed (Participants) | 68 | 51
score on a scale | 4.28 (8.13) | 1.65 (7.03)

8. Secondary Outcome: Change in Fitbit-measured Physical Activity Level
Description: Change in total daily step count as measured by Fitbit. Scores could range from 0 steps per day to over 20,000 steps per day. Higher scores reflect more steps per day.
Time Frame: assessed at baseline, 1, 2, 3, 4, 5, 6, 7, 8, 21 weeks; change from baseline to 21 weeks reported.
Population: 31 participants had useable data at baseline and 21 weeks. Fitbits were only added at the San Diego site.
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | ME-CCT | Supportive Contact Control Group
Number analyzed (Participants) | 16 | 15
steps | 146.62 (1962.36) | -867.84 (1198.58)

9. Secondary Outcome: Change in Fitbit-measured Sleep Time
Description: Change in total sleep time in minutes, per 24 hours, as measured by Fitbit. Possible scores range from 0-1440 (the number of minutes in 24 hours). Higher scores reflect more minutes of sleep.
Time Frame: assessed at baseline, 1, 2, 3, 4, 5, 6, 7, 8, 21 weeks; change from baseline to 21 weeks reported.
Population: 25 participants had useable data at baseline and 21 weeks. Fitbits were only used at the San Diego site.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ME-CCT Group | Supportive Contact Control Group
Number analyzed (Participants) | 12 | 13
minutes | -25.63 (90.29) | 11.57 (64.73)

ADVERSE EVENTS:
Time Frame: 21-week study
Description: No adverse events linked to study procedures.
Arm/Group | ME-CCT | Supportive Contact Control Group
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/66
Serious Adverse Events (participants affected / at risk) | 3/79 | 3/66
Other Adverse Events (participants affected / at risk) | 0/79 | 0/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ME-CCT (N=79) | Supportive Contact Control Group (N=66)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) — Hospitalized for urinary retention unrelated to study participation.
Slow heartbeat (Cardiac disorders) | 0 (0) | 1 (1) — Hospitalized for slow heartbeat due to medication overuse unrelated to study participation.
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) — Hospitalized for suicide attempt in the context of alcohol intoxication unrelated to study participation.
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) — Hospitalization for pneumonia unrelated to study participation.
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Hospitalization for COPD exacerbation unrelated to study participation.
COVID (Infections and infestations) | 0 (0) | 1 (1) — Hospitalization due to COVID infection unrelated to study participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT03225482/Prot_SAP_ICF_000.pdf